CLINICAL TRIAL: NCT03101917
Title: Microtable® Microstereotactic Frame and Drill Press and Associated Method for Cochlear Implantation
Brief Title: Microtable® Method for Cochlear Implantation Investigational Device Exemption (IDE)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Robert Labadie, Professor and Chair, Dept of O-HNS, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161659
Record Dates: First submitted 2017-03-15; First posted 2017-04-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Hearing Loss, Cochlear
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: All patients who meet eligibility requirements and choose to participate will undergo the image guided surgical cochlear implantation procedure as described in the protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Visual assessment of electrode insertion (Experimental): This arm will include the first 6 participants. In this group, a cut will be made near the eardrum and it will be lifted up so the surgeon can see the electrode as it goes into the cochlea.
  Interventions: Device: The Microtable® Stereotactic System
- Camera assessment of electrode insertion (Experimental): This arm will include the next 6 participants. In this group, a tube with a camera will be inserted past the ear drum, by making a small hole in the ear drum, to see the electrode as it goes into the cochlea.
  Interventions: Device: The Microtable® Stereotactic System

INTERVENTIONS:
Device: The Microtable® Stereotactic System — x

SUMMARY:
The Microtable® Microstereotactic Frame and Drill Press and Associated Method for Cochlear Implantation consists of a patient-customized microstereotactic frame which targets the cochlea. The intended use of the device in this early feasibility study is to surgically access the cochlea, allowing placement of an intra-cochlear electrode array for cochlear implantation, thereby providing a less invasive surgical option than currently performed. Compared to traditional cochlear implantation (CI) surgery, the investigators hypothesize that the minimally invasive, image-guided approach may offer the following benefits: (1) shorter procedure time including shorter general anesthesia time, (2) less tissue removal potentially eliminating post-operative mastoid bone depression, decreased post-operative patient discomfort, and quicker wound healing, (3) better chance of preservation of taste secondary to preservation of the chorda tympani nerve, and (4) standardization of electrode placement potentially allowing more consistent placement within the scala tympani sub-compartment of the cochlea which has been shown to be associated with improved post-operative audiological performance. This early feasibility study will focus on the advantages of the new technology to the patient. Advantages to the healthcare delivery system will be examined during the pivotal study phase.

DETAILED DESCRIPTION:
The Microtable® Microstereotactic Frame and Drill Press and Associated Method for Cochlear Implantation consists of a patient-customized microstereotactic frame which targets the cochlea. The intended use of the device in this early feasibility study is to surgically access the cochlea, allowing placement of an intra-cochlear electrode array for cochlear implantation, thereby providing a less invasive surgical option than currently performed. Compared to traditional cochlear implantation (CI) surgery, the investigators hypothesize that the minimally invasive, image-guided approach may offer the following benefits: (1) shorter procedure time including shorter general anesthesia time, (2) less tissue removal potentially eliminating post-operative mastoid bone depression, decreased post-operative patient discomfort, and quicker wound healing, (3) better chance of preservation of taste secondary to preservation of the chorda tympani nerve, and (4) standardization of electrode placement potentially allowing more consistent placement within the scala tympani sub-compartment of the cochlea which has been shown to be associated with improved post-operative audiological performance. This early feasibility study will focus on the advantages of the new technology to the patient. Advantages to the healthcare delivery system will be examined during the pivotal study phase.

The investigators propose this early feasibility study to determine if minimally invasive image-guided drilling to surgically access the cochlea for CI can be successfully performed. The study will involve only unilateral CI. The decision of unilateral vs. bilateral implantation is made clinically and before the patient may elect to enroll in this study. Bilateral implantation can take place either simultaneously or sequentially, with the decision made by the clinician as part of standard care.

If a participant is scheduled for routine bilateral CI, the traditional approach will be used on one side and the investigational approach on the other. Traditional surgery will be performed on the better-hearing ear, and the investigational technique will be performed on the poorer hearing ear. To minimize patient variability, the investigators will only be studying lateral wall electrodes, the Cochlear slim straight electrode and MED-EL electrodes. The investigators plan to enroll 12 cochlear implant patients in two groups. Group 1 will consist of patients implanted under direct visualization afforded by lifting a tympanomeatal flap, and Group 2 will consist of patients implanted with visualization afforded by passing an endoscope across the eardrum via a myringotomy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 22 to 80 years of age.
* Able to complete study related procedures.
* Able to provide written informed consent.
* Eligible for cochlear implant surgery as per routine pre-operative CI evaluation/workup. If patient is a candidate for bilateral CI, the research technique will be performed unilaterally on the side with the most favorable anatomy and/or worst residual hearing.
* Pre-operative CT scan of head/temporal bone as part of routine care showing normal temporal bone and intra-cochlear anatomy.
* Scheduled to receive either a Cochlear CI522 with the slim straight electrode or a MED-EL Synchrony with standard, Flex 24, or Flex 28 electrode.

Exclusion Criteria:

* Females who are pregnant. As part of routine pre-operative care, all females of childbearing potential will undergo either urine or blood pregnancy testing.
* ASA (American Society of Anesthesiologists) Physical Status classification of 4 or above or determined by surgeon to be too great of a health risk.
* Previous mastoidectomy on the ear undergoing research procedures.
* Severe anatomical abnormality of the temporal bone including but not limited to: 1) Mondini malformation 2) common cavity malformation 3) enlarged vestibular aqueducts (EVA) and/or 4) cochlea ossification.
* Severe chronic ear disease.
* Active middle ear infection.
* Subjects without a favorable trajectory based on pre-operative imaging, analysis and planning with favorable trajectory defined as a linear track extending from the surface of the mastoid cortex, through the facial recess, and targeting the basal turn of the cochlea without violation of the external auditory canal, sigmoid sinus, tegmen, and/or facial nerve.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-07-05 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Successful insertion of the CI electrode array into the cochlea. | Intraoperative
  Assessed by CT confirmation of intra-cochlear placement of the electrode array.

SECONDARY OUTCOMES:
Time in minutes of cochlear implant surgery. | immediately post-operative
  Assessed by physical exam immediately after surgical intervention.
Amount of tissue removed scanning | pre-operative and post-operative
  Volume assessed by comparison of pre-operative CT scan to the post-operative CT scan
Preservation of taste scanning | 2-4 weeks post-operative
  Assessed by postoperative survey
Optimal electrode position within the cochlea's scala tympani scanning | Intraoperative
  Assessed by intraoperative CT scan
Avoidance of damage to the facial nerve during the image guided cochlear implantation surgery. | up to 12 months post-operative
  Assessed by physical exam immediately after surgical intervention and follow-up visits via the House-Brackmann scale.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Labadie, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No